CLINICAL TRIAL: NCT00695448
Title: A Phase I Open-Label, Dose-Escalation Study of the Phosphoinositide 3-Kinase Inhibitor GSK1059615 in Patients With Solid Tumors or Lymphoma
Brief Title: Phase I Open-Label, Dose-Escalation Study of GSK1059615 in Patients With Solid Tumors or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated prematurely due to lack of sufficient exposure following single- and repeat-dosing.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIK111051
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Solid Tumours
Keywords: Phosphoinositide 3-kinase inhibitor; solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohorts (Experimental): The starting dose is 6mg once daily (QD); dose is to be escalated using a standard 3 + 3 dose escalation scheme.
  Interventions: Drug: GSK1059615

INTERVENTIONS:
Drug: GSK1059615 — GSK1059615 is dosed orally once daily for 21 days of a 28-day cycle. Patients continue treatment for subsequent cycles as long as eligible and receiving benefit.

SUMMARY:
This is an open-label, multi-center Phase I study conducted to define the recommended Phase 2 dose, toxicity profile, pharmacokinetics and biologically active dose range of GSK1059615.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* 18 years old or older.
* Histologically- or cytologically- confirmed diagnosis of solid tumor malignancy or lymphoma that is not responsive to accepted standard therapies or for which there is no standard or curative therapy.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* A life expectancy of > 12 weeks.
* Able to swallow and retain oral medication.
* A male is eligible to enter and participate in the study if he either:
* agrees to abstain from sexual intercourse from the first dose of study drug and until 21 days after last dose of study medication, or
* agrees to use a condom and occlusive cap (diaphragm or cervical/vault cap) with spermicidal foam/gel/film/cream/suppository from the first dose of study drug and until 21 days after last dose of study medication, or
* is surgically sterile. NOTE: Male patients must use contraception to prevent pregnancy in a female partner and prevent exposure of any partner to semen by any means (refer to protocol).
* A female is eligible to enroll in the study if she is of:

Non-child bearing potential (i.e., physiologically incapable of becoming pregnant) including any woman who is characterized by at least one of the following:

* Has had a hysterectomy
* Has had a bilateral oophorectomy (ovariectomy)
* Has had a bilateral tubal ligation
* Is post-menopausal (total cessation of menses for ≥ 1 year) Childbearing potential, has a negative serum pregnancy test at screening, and agrees to one of the following from at least 2 weeks prior to the first dose of study drug and until 21 days after last dose of study medication:
* Use an intrauterine device (IUD) with a documented failure rate of
* less than 1% per year.
* Have intercourse only with a vasectomized partner who is sterile
* and is the sole sexual partner for that woman.
* Complete abstinence from sexual intercourse.
* Use double barrier contraception defined as condom with
* spermicidal jelly, foam, suppository, or film; OR diaphragm with
* spermicide; OR male condom and diaphragm. NOTE: Oral contraceptives are not reliable due to potential for drug-drug interaction.
* Adequate organ system function as defined in the protocol.

Exclusion Criteria:

* Use of an investigational anti-cancer drug within 28 days or 5 half-lives preceding the first dose of GSK1059615.
* Chemotherapy within the last 3 weeks (6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity are permitted with approval of the GSK medical monitor if administered at least 2 weeks prior to the first dose of study drug.
* Trastuzumab within the last 4 weeks.
* Any major surgery, radiotherapy, or immunotherapy within the last 4 weeks.
* Prior use of any PI3K inhibitor.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug. (To date there are no known FDA approved drugs chemically related to GSK1059615).
* Current use of a prohibited medication or requires any of these medications during treatment with GSK1059615 as per protocol.
* Current use of warfarin for therapeutic anticoagulation.
* NOTE: Low molecular weight heparin and prophylactic low-dose warfarin are permitted. PT/PTT must meet the inclusion criteria. Patients taking warfarin must have their INR followed closely.
* Presence of an active gastrointestinal disease or other condition known to interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
* Unresolved toxicity greater than Grade 1 from previous anti-cancer therapy except alopecia. Patients with stable Grade 2 neuropathy can be enrolled with approval by the GSK Medical Monitor.
* QTc interval ≥ 480 msecs.
* History of acute coronary syndromes (including unstable angina and myocardial infarction), atrial fibrillation, coronary angioplasty, or stenting within the past 24 weeks.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Symptomatic or untreated leptomeningeal or brain metastases. Patients previously treated for these conditions who are asymptomatic and off of corticosteroid and P450-inducing anti-epileptic medication for at least 2 months are permitted.
* Primary malignancy of the central nervous system.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
* Nursing female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-06-24 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) and changes in laboratory values and vital signs as per protocol. | 21 days

SECONDARY OUTCOMES:
Pharmacokinetic parameter values for GSK1059615 following single and repeated dosing, including area under the plasma drug concentration curve (AUC), maximum observed plasma drug concentration (Cmax) | 21 days
time to maximum observed plasma drug concentration, and half-life of GSK1059615. | 21 days
Metabolic profiling in plasma and urine, and amount excreted in urine (subset of patients). | 21 days
Tumor response as defined by RECIST in the protocol. | 56 days
Change from baseline in protein markers in tumor and/or blood. | 28 days
Blood glucose and insulin levels. | Daily for 28 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: PIK111051 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: PIK111051 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: PIK111051 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: PIK111051 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: PIK111051 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: PIK111051 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: PIK111051 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register